CLINICAL TRIAL: NCT01685723
Title: Helping Cancer Patients Quit Smoking Using Brief Advice Based on Risk Communication: a Randomized Controlled Trial
Brief Title: Smoking Cessation in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Food and Health Bureau, Hong Kong (Other Government); Queen Mary Hospital, Hong Kong (Other); Tuen Mun Hospital (Other Government); Queen Elizabeth Hospital, Hong Kong (Other); Princess Margaret Hospital, Hong Kong (Other Government); Pamela Youde Nethersole Eastern Hospital (Other)
Responsible Party: Principal Investigator, Prof. Sophia Siu-chee Chan, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: cancer_rct_1
Record Dates: First submitted 2012-08-26; First posted 2012-09-14 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Cancer; Smoking Cessation
Keywords: Cancer patients; Smoking cessation; Risk communication
MeSH Terms: conditions — Neoplasms; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Counseling group (Experimental): Subjects in this group will receive a face-to-face individualized brief advice based on risk communication for 15-30 minutes from the nurse counselors and a booster intervention (10-15 minutes) at 1 week.
  Data collection will be conducted at 1 week, 1, 3, 6, 9, 12 months via telephone.Ten subjects from the intervention group who have not quitted will be invited for a process evaluation in the form of face-to-face interviews by research assistants at 12-month follow-up.
  Interventions: Behavioral: Counseling group
- General supporting (Sham Comparator): Subjects in this group will receive standard care without risk communication.
  Data collection will be conducted at 1 week, 1, 3, 6, 9, 12 months via telephone.
  Interventions: Behavioral: General supporting

INTERVENTIONS:
Behavioral: Counseling group — Subjects will receive brief advice based on risk communication by a nurse counselor. The brief advice will be based on a specifically-designed risk communication leaflet that warns about the risks of continued smoking for subjects' cancer treatment and prognosis. Subjects will receive a booster intervention via telephone at 1 week to assess the progress of and barriers to the subjects' action plans and identifying individual difficulties and facilitators towards quitting. They also receive a generic standard self-help smoking cessation booklet.
  Arms: Counseling group
Behavioral: General supporting — Subjects in this group will receive a generic self-help smoking cessation booklet and standard care without risk communication. They will have the same follow-up sections as the intervention group to receive diseases support.
  Arms: General supporting

SUMMARY:
Background: Smoking cessation can largely improve cancer prognosis and quality of life among cancer patients. However, few patients are aware of the importance to quit at the stage, or they have difficulties to quit by self.

Aim: to examine the effectiveness of a smoking cessation intervention using a risk communication approach

Design: A randomized controlled trial

Setting: Outpatient clinics of the Clinical Oncology Departments of five major hospitals in different regions of Hong Kong

Subject: Smokers who attend medical follow-up visits at outpatient clinics of the Clinical Oncology Departments of five major hospitals in different regions of Hong Kong and who met the inclusion criteria were invited to participate.

Intervention: At baseline, intervention group receives:

1. a face-to-face individualized brief advice based on risk communication for 15-30 minutes from the nurse counselors;
2. examination of exhale CO level; and
3. a generic standard self-help smoking cessation booklet. They will receive a booster intervention at 1 week. Control group will receive standard care and a generic self-help smoking cessation booklet.

Outcome: Primary outcome is the self-reported 7-day point prevalence quit rate at 6-month follow up. Secondary outcomes include:

1. self-reported 7-day point-prevalence smoking abstinence at 12-month follow-up;
2. biochemically validated quit rate at 6-month follow-up; and
3. percentage of patients reduced smoking by at least 50% at 6- and 12-month follow-up compared to baseline.

Significance: This study develops and validates practical smoking cessation interventions targeted to cancer patients to improve their cancer prognosis and in long-term.

DETAILED DESCRIPTION:
Smoking causes many types of cancer in general. Past studies have shown that current smokers have increased risk of cancer, and most lung cancers are attributable to smoking. Cancer (malignant neoplasm) is the number one killer in Hong Kong, which leads to nearly one-third of all deaths each year. Cancer patients who continue smoking would result in extra risks of all cause mortality, cancer recurrence and second primary cancer as well as reducing survival time (Chen et al., 2010). Smoking could also reduce the efficacy of clinical and medical treatment of cancer including radio- and chemo-therapies (Benninger et al., 1994; Browman et al., 1993) and increase the risk of treatment related side-effects (Rugg et al., 1990).

Cancer patients may present an excellent "teachable moment" for smoking cessation interventions, as their current illness could largely be due to smoking. However, few smoking cessation programs target on this vulnerable group and only one-third of oncology nurses would assist cancer patients quit smoking. Healthcare professionals have the responsibility to assist this vulnerable group to quit smoking. Recent randomized controlled trials (RCT) suggested behavioral intervention may help cancer patients quit smoking, but they are limited by small sample size. No RCT study has ever been done in Hong Kong.

This study can make an important contribution to evidence-based practice by testing the effectiveness of a smoking cessation intervention using a risk communication approach and targeting cancer patients. The results primarily serve the purpose to support the development of clinical practice guidelines and interventions to promote smoking cessation in cancer patients to improve their cancer prognosis and, in the long-run, increase their survival time and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* patients smoked at least weekly in the past 6 months;
* diagnosed with cancer not limited to smoking-induced cancers;
* patients in all stages 0,I,II,III, or IV;
* aged 18 or above; and
* can communicate in Cantonese

Exclusion Criteria:

* those with unstable medical conditions as advised by the doctor in charge;
* poor cognitive state or with mental illness; and
* those participating in other smoking cessation program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The self-reported 7-day point prevalence (pp) quit rate at 6 months | 6 months
  Whether the participant has quitted smoking in the past seven days at the time point of 6 months

SECONDARY OUTCOMES:
The self-reported 7-day point prevalence (pp) quit rate at 12 months | 12 months
  Whether the participant has quitted smoking in the past seven days at the time point of 12 months
Biochemical validation of smoking status at 6 months | 6 months
  Biochemically validated quit rate (saliva cotinine level and exhale CO test)
Percentage of patients reduced smoking by at least 50% at 6 months | Baseline and 6 months
  Percentage of patients reduced smoking by at least 50% at 6 months
Percentage of patients reduced smoking by at least 50% at 12 months | Baseline and 12 months
  Percentage of patients reduced smoking by at least 50% at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sophia SC Chan, PhD, MPH, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China

REFERENCES:
- [Background] Benninger MS, Gillen J, Thieme P, Jacobson B, Dragovich J. Factors associated with recurrence and voice quality following radiation therapy for T1 and T2 glottic carcinomas. Laryngoscope. 1994 Mar;104(3 Pt 1):294-8. doi: 10.1288/00005537-199403000-00009. PMID 8127185
- [Background] Browman GP, Wong G, Hodson I, Sathya J, Russell R, McAlpine L, Skingley P, Levine MN. Influence of cigarette smoking on the efficacy of radiation therapy in head and neck cancer. N Engl J Med. 1993 Jan 21;328(3):159-63. doi: 10.1056/NEJM199301213280302. PMID 8417381
- [Background] Rugg T, Saunders MI, Dische S. Smoking and mucosal reactions to radiotherapy. Br J Radiol. 1990 Jul;63(751):554-6. doi: 10.1259/0007-1285-63-751-554. PMID 2390690
- [Background] Chen J, Jiang R, Garces YI, Jatoi A, Stoddard SM, Sun Z, Marks RS, Liu Y, Yang P. Prognostic factors for limited-stage small cell lung cancer: a study of 284 patients. Lung Cancer. 2010 Feb;67(2):221-6. doi: 10.1016/j.lungcan.2009.04.006. Epub 2009 Jun 3. PMID 19497635
- [Derived] Li WH, Chan SS, Wang KM, Lam TH. Helping cancer patients quit smoking by increasing their risk perception: a study protocol of a cluster randomized controlled trial. BMC Cancer. 2015 Jun 30;15:490. doi: 10.1186/s12885-015-1496-2. PMID 26122078